CLINICAL TRIAL: NCT04397250
Title: The Effect of High-intensity Interval Training on Biomarkers of Cardiometabolic Health in Persons With Chronic Paraplegia: A Randomised Controlled Trial
Brief Title: High-intensity Interval Training for Cardiometabolic Health in Persons With Spinal Cord Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Bath (Other)
Responsible Party: Principal Investigator, James Bilzon, Professor, University of Bath
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20/SW/0051
Record Dates: First submitted 2020-05-17; First posted 2020-05-21 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Paraplegia
Keywords: high-intensity interval training; cardiometabolic health
MeSH Terms: conditions — Paraplegia | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity interval training (Experimental): Participants will be asked to perform four 30 minutes bouts of high-intensity interval exercise per week.
  Interventions: Behavioral: High-intensity interval training
- Control (No Intervention): Participants will be asked to continue their habitual lifestyle

INTERVENTIONS:
Behavioral: High-intensity interval training — Arm-cranking exercise
  Arms: High-intensity interval training

SUMMARY:
Persons with chronic paraplegia at an increased risk of developing cardiovascular disease and type-2 diabetes compared to the able-bodied population. There is mounting evidence from the able-bodied literature that high-intensity interval training (HIIT) is an effective way to improve cardiometabolic health outcomes, but this effect has yet to be investigated in persons with chronic paraplegia.

This study is recruiting adults (aged 18-65 years) with paraplegia (T2 or below) who sustained their spinal cord injury more than one-year ago. Participants will need to attend the laboratory at the University of Bath on two occasions (baseline and follow-up testing) separated by eight weeks. Following the first visit, participants will be randomised to a exercise group or control group. For those in the exercise group, participants will be provided with an arm crank ergometer for use in their home, and be asked to perform four exercise sessions per week (30 min each) for six weeks. For those in the control group, participants will be asked to continue their normal lifestyle.

DETAILED DESCRIPTION:
The aim of this research is to determine the effect of HIIT (vs. a control group) on biomarkers of cardiometabolic health in persons with chronic paraplegia.

Baseline and follow-up assessments:

Before each visits, participants will be asked to refrain from any strenuous physical activity (2 days prior), consume no caffeine (including tea or coffee) or alcohol (1 day prior), and have fasted for at least 10 hours overnight before arriving to the University of Bath laboratories.

There will be measurements of basic anthropometrics (height, weight, waist and hip circumference), body composition (via a DEXA scan), resting metabolic rate, sub-maximal and maximal exercise capacity, and blood responses following the consumption of a sugary drink.

Physical activity and diet monitoring:

Participants will be asked to monitor their normal diet (weighed food diary) and physical activity patterns (chest-worn strap) over a 1-week period following the first visit, and in the final week of the 6-week intervention/control period.

Exercise intervention:

The 6-week exercise programme or control will start two weeks after the first lab visit. Participants in the exercise group will be asked to wear a heart-rate monitor for all exercise sessions, and upload their data to a smartphone for remote-monitoring by the research team.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a chronic (>12 months post-injury) SCI below T2
* Individuals who spend >75% of their waking day in a wheelchair
* Weight stable (weight not changed by >3% over the last 3 months)

Exclusion Criteria:

* Individuals who an acute (<12 months post-injury) SCI
* Individuals who spend <75% of their waking day in a wheelchair
* Individuals on type-2 diabetes medication
* Individuals self-reporting active medical issues (pressure sores, urinary tract infections, cardiac disorders, musculoskeletal complaints of the upper extremities, or cardiovascular contraindications to exercise testing)
* Plans to change lifestyle during the study period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Fasting insulin | 6 weeks
  Serum insulin concentration
Peak aerobic capacity | 6 weeks
  Measured using a incremental ramp protocol on a arm crank ergometer
Peak power output | 6 weeks
  Maximum power output achieved during peak aerobic capacity test

SECONDARY OUTCOMES:
Body mass | 6 weeks
  Measured using electronic wheelchair scales
Waist and hip circumference | 6 weeks
  Measured using a non-metallic tape
Total body fat percentage | 6 weeks
  Measured using duel-energy x-ray absorptiometry
Total Fat Mass | 6 weeks
  Measured using duel-energy x-ray absorptiometry
Total Fat-Free Mass | 6 weeks
  Measured using duel-energy x-ray absorptiometry
Visceral Adipose Tissue | 6 weeks
  Measured using duel-energy x-ray absorptiometry
Systolic and diastolic blood pressure | 6 weeks
  Measuring using a automated sphygmomanometer
Resting metabolic rate | 6 weeks
  Measured using indirect calorimetry
Time spent in different physical activity intensities (MET categories) (minutes) | 6 weeks
  Time spent in different physical activity intensities across 7-days (MET categories) (minutes)
Energy expended in different physical activity intensities (MET categories) (kJ or kcal) | 6 weeks
  Energy expended in different physical activity intensities across 7-days (MET categories) (kJ or kcal)
Energy intake and dietary macronutrient composition | 6 weeks
  Estimated using a 7-day weighed food diary
Fasting metabolite/hormone/inflammatory profile | 6 weeks
  Assessment of blood glucose, glycated hemoglobin, triglycerides, non-esterified fatty acids, total cholesterol, high density lipoprotein, and low density lipoprotein concentrations, leptin, C-reactive protein, interleukin-6, tumour-necrosis factor-alpha, and adiponectin
Postprandial metabolites | 6 weeks
  Assessment of blood glucose and insulin
Shoulder Pain | 6 weeks
  Measured using a validated questionnaire
Exercise Self-Efficacy | 6 weeks
  Measuring using a validated questionnaire
Health-related quality of life | 6 weeks
  Measured using a validated questionnaire
Fatigue | 6 weeks
  Measured using a validated questionnaire
Independence | 6 weeks
  Measured using a validated questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: James Bizon, Principal Investigator — University of Bath
Locations (1):
- University of Bath, Bath, United Kingdom

REFERENCES:
- [Derived] Farrow MT, Maher J, Thompson D, Bilzon JLJ. Effect of high-intensity interval training on cardiometabolic component risks in persons with paraplegia: Protocol for a randomized controlled trial. Exp Physiol. 2021 May;106(5):1159-1165. doi: 10.1113/EP089110. Epub 2021 Mar 20. PMID 33600014